CLINICAL TRIAL: NCT01928784
Title: Radial Extracorporeal Shock Wave Therapy on Chronic Low Back Pain: a Prospective Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Cheng Zeng, MD, Beijing Jishuitan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SW-LBP-01
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Low Back Pain
Keywords: Low back pain; extracorporeal shock wave therapy; Trigger Points
MeSH Terms: conditions — Low Back Pain | interventions — Emergency Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Specific pain spot (Experimental): Radial Extracorporeal Shock Wave Therapy 2000 impulses, Patients with specific pain spot for low back pain
  Interventions: Device: Radial Extracorporeal Shock Wave Therapy 2000 impulses
- No specific pain spot (Experimental): Radial Extracorporeal Shock Wave Therapy 4000 impulses, Patients without specific pain spot for low back pain
  Interventions: Device: Radial Extracorporeal Shock Wave Therapy 4000 impulses

INTERVENTIONS:
Device: Radial Extracorporeal Shock Wave Therapy 2000 impulses — Radial Extracorporeal Shock Wave Therapy, 13 Hz, 2.5 Bar, 2000 impulses
  Other Names: SWISS DOLORCLAST® CLASSIC, EMS, Swiss
  Arms: Specific pain spot
Device: Radial Extracorporeal Shock Wave Therapy 4000 impulses — Radial Extracorporeal Shock Wave Therapy, 13 Hz, 2.5 Bar, 4000 impulses
  Other Names: SWISS DOLORCLAST® CLASSIC, EMS, Swiss
  Arms: No specific pain spot

SUMMARY:
The aim of this prospective study is to explore the pain-alleviating effect of low-energy extracorporeal shock wave therapy(ESWT) in patients with chronic low back pain.

DETAILED DESCRIPTION:
26 patients who suffered from persistent symptoms for more than 3 months are going to be treated with DOLORCLAST radial extracorporeal shock wave(EMS, Swiss). Patients are assigned to two groups according to the exist of specific pain spot. Group I(have specific pain spot) received a total of 2000 impulses of 2.5 Bar; group II(controls, no specific pain spot) 4000 impulses of 2.5 Bar. Patients is going to be treated once. The efficacy of therapy is going to be evaluated by VAS scale before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptom of low back pain during last 4 weeks
* Low back pain history for more than 3 months

Exclusion Criteria:

* Have lower limbs radiating pain beyond knee joints
* Spinal tumorous or infectious disease, fracture, ankylosing spondylitis, cauda equina syndrome or other severe spinal diseases
* Spinal surgical history
* Severe heart, lung, liver, kidney disease or high blood pressure
* With cardiac pacemaker
* Coagulopathy or thrombosis
* Have ESW therapy or pharmaceutical treatment for low back pain during last 1 months
* Mental illnesses or none cooperation
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Change in Visual analogue scale scores(VAS) of patients before and after therapy | baseline, 1 hour after therapy
  Change of Visual analogue scale score(VAS) of patients before and after shock wave therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yajun Liu, MD, Study Director — Beijing Jishuitan Hospital; Yan An, MD, Principal Investigator — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Dagenais S, Tricco AC, Haldeman S. Synthesis of recommendations for the assessment and management of low back pain from recent clinical practice guidelines. Spine J. 2010 Jun;10(6):514-29. doi: 10.1016/j.spinee.2010.03.032. PMID 20494814